CLINICAL TRIAL: NCT02976467
Title: A Randomized, Double-blind, Multicenter Study to Assess the Safety and Efficacy of a 6 Month Oral Treatment With the Chymase Inhibitor BAY 1142524 at a Dose of 25 mg BID in Comparison to Placebo on Top of Standard of Care in Patients With Reduced Left-ventricular Ejection Fraction (LVEF≤ 45%) After Acute Myocardial Infarction
Brief Title: A Double-blind Study to Investigate Efficacy, Safety and Tolerability of BAY 1142524 in Patients After Acute Myocardial Infarction With Left-ventricular Dysfunction
Acronym: CHIARA MIA 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16673; 2016-002167-33 (EudraCT Number)
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — fulacimstat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fulacimstat (BAY1142524) (Experimental): 30 patients with left-ventricular dysfunction after acute myocardial infarction
  Interventions: Drug: Fulacimstat (BAY1142524)
- Placebo (Placebo Comparator): 30 patients with left-ventricular dysfunction after acute myocardial infarction
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fulacimstat (BAY1142524) — 25 mg BAY 1142524 are given twice daily over a treatment period of 6 months
  Arms: Fulacimstat (BAY1142524)
Drug: Placebo — Matching placebo tablets are given twice daily over a treatment period of 6 months
  Arms: Placebo

SUMMARY:
The purpose of the trial is the analysis of safety and efficacy of the chymase inhibitor BAY1142524 at a dose of 25 mg BID in comparison to placebo using a 6 months treatment period in patients with left-ventricular (LV) dysfunction after myocardial infarction (MI). BAY1142524 or placebo will be given on top of evidence-based standard of care for left-ventricular dysfunction after myocardial infarction. Primary objective is the analysis of first signs of efficacy as determined by favourable changes in functional parameters of adverse cardiac remodelling (i.e. endsystolic and enddiastolic volume index, ejection fraction). Secondary objective is the analysis of safety and tolerability as evidenced by the incidence and severity of adverse events. 30 patients have to complete treatment with verum and 30 patients have to complete treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first ST elevation myocardial infarction (STEMI) treated with primary percutaneous intervention (PCI) or thrombolysis within 24 hours after symptom onset
* Diagnosis of STEMI requires the presence of the following three criteria:

  * Typical clinical symptoms such as chest pain, shortness of breath for more than 20 minutes related to the myocardial infarction
  * New ST elevation indicating myocardial infarction
  * Significant elevation in troponin T or I with at least one value above the 99th percentile upper reference limit (URL) and/or elevation creatine kinase (CK) and creatine kinase MB (6-10% of total CK)
* At the screening period, on day 5 to 9 after MI, patients have to have a LVEF ≤ 45% and an infarct size >10% LV mass (as measured by LGE-MRI, central-blinded evaluation)

Exclusion Criteria:

* Contraindication to perform contrast-enhanced cardiac MRI
* LVEF < 20%
* History of heart failure or LVEF < 50% before occurrence of the first STEMI
* Infarct size > 45% (g/g; LV mass) between 5 and 9 days after myocardial infarction
* NYHA (New York Heart Association) class IV at randomization
* Any planned cardiac intervention after baseline MRI or any other planned operations
* Non-ischemic causes for cardiomyopathy
* Diagnosis of atrial fibrillation
* Systolic blood pressure < 100 mm Hg or > 180 mm Hg; diastolic blood pressure < 50 mm Hg or >110 mm Hg, heart rate < 50 or >100 beat/minute; mean of triplicate values at randomization
* Clinically relevant hepatic dysfunction

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Change in left-ventricular ejection fraction (LVEF) | At 6 months
Change in end diastolic volume index (EDVI) | At 6 months
Change in end systolic volume index (ESVI) | At 6 months

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to 7 months
Number of patients with serious adverse events | Up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- Czechia (2):
  - Kladno
  - Prague
- Germany (4):
  - Hanover, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Erfurt, Thuringia
  - Berlin
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (4):
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Milan, Lombardy
  - Monza-Brianza, Lombardy
- Spain (4):
  - Babio - Beade, Pontevedra
  - Barcelona
  - Madrid
  - Valencia

REFERENCES:
- [Derived] Duengen HD, Kim RJ, Zahger D, Orvin K, Kornowski R, Admon D, Kettner J, Shimony A, Otto C, Becka M, Kanefendt F, Romo AI, Hasin T, Ostadal P, Rojas GC, Senni M; GROUP investigators of the CHIARA MIA 2 trial. Effects of the chymase inhibitor fulacimstat on adverse cardiac remodeling after acute myocardial infarction-Results of the Chymase Inhibitor in Adverse Remodeling after Myocardial Infarction (CHIARA MIA) 2 trial. Am Heart J. 2020 Jun;224:129-137. doi: 10.1016/j.ahj.2020.01.012. Epub 2020 Jan 25. PMID 32375104